CLINICAL TRIAL: NCT05792202
Title: Combined Microfracture Procedure Promotes Tendon Healing During Double Raw Repair for Full Tear Rotator Cuff - a Prospective Randomized Study With 2-year Follow-up
Brief Title: Combined Microfracture Procedure Promotes Tendon Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Yi Lu, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY
Record Dates: First submitted 2023-03-18; First posted 2023-03-31 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Full Rotator Cuff Tear; Microfracture Procedure; Double Raw Repair

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): double raw repair for full tear rotator cuff combined microfracture procedure
  Interventions: Procedure: microfracture procedure
- Control group (Placebo Comparator): double raw repair for full tear rotator cuff
  Interventions: Procedure: only double raw repair

INTERVENTIONS:
Procedure: microfracture procedure — double raw repair combined with microfracture procedure which promotes tendon healing by releasing growth factors
  Arms: Study group
Procedure: only double raw repair — the double raw repair was used to repair the tendon tear
  Arms: Control group

SUMMARY:
This study is a prospective randomized controlled study of Combined microfracture procedure promotes tendon healing during double raw repair for full tear rotator cuff. The patients with rotator cuff tear were randomly divided into groups before the operation. The patients were followed up before and 6 weeks, 3 months, 6 months, 12 months after surgery. In different time periods, the quantitative and qualitative indicators including pain, functional score, muscle strength, MRI performance, etc. were compared between groups at the same time period to evaluate the difference in the effect of Crimson duvet procedure with Greenhouse procedure on the treatment of rotator cuff.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopy confirmed small to medium full rotator cuff tear
* Unilateral rotator cuff injury
* Voluntarily accept randomized controlled grouping, cooperate with treatment and follow up patients
* Young and middle-aged patients aged 20 to 60

Exclusion Criteria:

* Previous shoulder surgery (incision or arthroscopy)
* Combined with diseases of other parts of the same limb
* Combined with Bankart injury, acromioclavicular joint disease, greater tuberosity fracture, glenoid fracture and so on
* Bilateral onset
* Unable or unwilling to receive clinical follow-up

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
rotator cuff re-tear rate | 2 year postoperatively
  the rotator cuff re-tear rate was measured by MRI, MRI was performed to identify the status of the tendon

SECONDARY OUTCOMES:
VAS (Visual Analogue Scale) | 1,2,3,7 days postoperatively and 3,6,12,24 months postoperatively, higher scores mean a worse outcome.
  A score used to evaluate the pain
ASES（American Shoulder and Elbow Surgeons'Form） | 3,6,12,24 months postoperatively
  A score used to evaluate the shoulder function, higher scores mean a better outcome.
Constant score | 3,6,12,24 months postoperatively
  A score used to evaluate the shoulder function, higher scores mean a better outcome.
UCLA (University LosAngeles scoring system) | 3,6,12,24 months postoperatively
  A score used to evaluate the shoulder function, higher scores mean a better outcome.
SST (simple shoulder test) | 3,6,12,24 months postoperatively
  A score used to evaluate the shoulder function, higher scores mean a better outcome.
front extension, external rotation and internal rotation strength of shoulder | 6,12,24 months postoperatively
  Use a dynamometer to measure in N

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No